CLINICAL TRIAL: NCT04741425
Title: Effects of an Online Theory-based Educational Programme for Primiparous Women on Improving Breastfeeding Related Outcomes: A Randomised Controlled Trial
Brief Title: Online Theory-based Educational Programme for Primiparous Women on Improving Breastfeeding Related Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, WONG Mei Sze, PhD candidate, registered nurse, registered midwife, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 2020.577
Record Dates: First submitted 2021-02-02; First posted 2021-02-05 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Breastfeeding, Exclusive; Self Efficacy
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Masking Description: The group allocation is determined by the recruitment sequence into the study. Sealed, opaque envelopes with random codes (A and B) in blocks will be generated by a research assistant, who is blinded to the study group to maintain the randomization concealment, and the participant list with the group allocation will be prepared by another research assistant.
  Outcome assessment will be blinded by using online questionnaires.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- REST intervention (Experimental): There will be one session of online antenatal breastfeeding talk, 5 sessions of daily online postnatal individualized breastfeeding coaching, and 7 weekly postnatal telephone follow-ups.
  Interventions: Other: REST intervention
- Usual care (No Intervention): Standard antenatal and postnatal care provided by midwives and lactation consultants in the hospitals through by Zoom or by online self-learning through watching videos and reading pamphlets. Participants can also attend other breastfeeding talks or breastfeeding support groups provided by the non-governmental organizations for maternal care.
  After delivery, mothers will be taught about baby care at bedside. Breastfeeding skills will also be taught and assessed by the midwives and lactation consultants individually or in group-based breastfeeding talk in the postnatal ward.
  Upon discharge, a breastfeeding and postnatal hotline will be provided to all women for advices, and a telephone follow-up will be arranged for all the mothers within 3 to 4 days after delivery by midwives or lactation consultants. The mother-baby dyads will be suggested to follow up in MCHCs for baby growth and breastfeeding support.

INTERVENTIONS:
Other: REST intervention — The breastfeeding talk will be conducted by Zoom at the third trimester about breastfeeding benefits and other practical advices. There is also a sharing session by a successful breastfeeding mother and a group discussion with different breastfeeding scenarios.
  Once the mothers return home after delivery, individualized breastfeeding coaching will be provided by PI through a daily Zoom videoconference within 24 hours upon hospital discharge till Day 7 after delivery.
  During the last breastfeeding videoconference, mothers will be reminded to have weekly telephone follow-ups by PI from week 2 to 2 months postpartum.
  Women who are randomised into the intervention group will receive REST in addition to the standard antenatal and postnatal care (described at below) by the Obstetrics Department of their delivery hospitals.
  Arms: REST intervention

SUMMARY:
Breastmilk is the best food for babies and exclusive breastfeeding is beneficial to mother-baby dyads.

It is recommended to exclusively breastfeed babies till 6 months of age and continue with complementary food until aged 2 or above. This proposed study aims to establish and evaluate an effective intervention in sustaining exclusive breastfeeding among primiparous women up to 6 months postpartum.

DETAILED DESCRIPTION:
World Health Organization suggests all infants should be exclusively breastfed for 6 months and continue with complementary food till 2 years old. Yet, the global exclusive breastfeeding rate at 6 months is only around 40%. As for Hong Kong, breastfeeding rate dropped substantially from 87% upon discharge to less than a half at 6 months postpartum and only one-third of women still exclusively breastfed their infants.

According to previous studies, women had early breastfeeding initiation or had breastfed their first child for at least 6 months were more likely to exclusively breastfeed the babies for longer time. However, mothers have early weaning easily due to inadequate breastfeeding knowledge/ skills, lack of lactation support or if they have specific characteristics like being hypertensive/ diabetic, primiparous or having complicated birthing experience. It was also found that maternal breastfeeding education, breastfeeding self-efficacy and their intention all affect the initiation and continuation of breastfeeding.

Among various promotional interventions, educational and supportive interventions were found to be effectively increased breastfeeding duration, while self-efficacy based intervention improved breastfeeding self-efficacy in the first 2 months but not on exclusive breastfeeding rates at 6 months postpartum. In addition, overall, there are inconsistent effects on educational and supportive interventions on breastfeeding outcomes, especially exclusive breastfeeding rate at 6 months postpartum. Also, most of the previous reviews did not focus on the primiparous women. And it is unclear the intervention effects on breastfeeding self-efficacy and exclusive breastfeeding rate of the first time mothers over 6-months.

As a result, a systematic review of 13 randomised controlled trials was done to identify effective approaches to educational and supportive interventions to improve breastfeeding in first time mothers up to at least 6-month postpartum. The result showed educational and supportive interventions were effective in increasing exclusive breastfeeding rate at ≤2 months & 6 months, partial breastfeeding rate as well as breastfeeding self-efficacy at ≤2 months. The key components in breastfeeding promotion interventions, are those involved multicomponent (that is antenatal group education, postnatal individual breastfeeding coaching together with telephone follow-ups), breastfeeding self-efficacy theory-based that delivered across antenatal and postnatal period with ≥ 3 intervention sessions.

With the current COVID-19 pandemic, all face-to-face interventions in the hospitals are constrained. So the proposed study will be conducted by using Zoom platform and telephone follow-ups. There are one session of online antenatal breastfeeding talk, 5 times daily online postnatal breastfeeding coaching and 7 times weekly postnatal telephone follow-ups. The intervention will be guided by Dennis's breastfeeding self-efficacy framework.

This study aims to determine if a real-time online theory-based education and support plus telephone follow-ups programme (REST) for primiparous women in Hong Kong would increase their exclusive rate, breastfeeding self-efficacy, and other breastfeeding outcomes over 6-month postpartum.

ELIGIBILITY:
Inclusion Criteria:

* Hong Kong Chinese residents
* at the third trimester (≥32 weeks of gestation)
* aged ≥18 years
* having singleton pregnancy
* able to understand and write in Chinese and speak Cantonese
* delivered in the local public hospitals
* have access to Internet and able to use computer, smartphone or tablet.

Exclusion Criteria:

* having serious medical or obstetric complications such as hypertension and/or diabetes
* having psychiatric illness such as depression or schizophrenia
* not staying in Hong Kong for at least 6 months post-delivery
* having complicated delivery (e.g., instrumental or operative delivery, and/or postpartum hemorrhage)
* receiving pharmacological pain relief during their labor
* having baby admitted to the hospital during the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Primiparous women
Enrollment: 190 (Actual)
Dates: Start 2021-02-09 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Exclusive breastfeeding rate (number of Infants who have only received breastmilk or expressed breastmilk, and no other liquids or solids except vitamins, mineral supplement and medicines) by self-developed postnatal questionnaires | At 2 months postpartum (immediately post-intervention)
  The self-developed postnatal questionnaires are reviewed and commented by 3 lactation consultants and 2 midwives and revised accordingly.
Exclusive breastfeeding rate (number of Infants who have only received breastmilk or expressed breastmilk, and no other liquids or solids except vitamins, mineral supplement and medicines) by self-developed postnatal questionnaires | At 6 months postpartum
  The self-developed postnatal questionnaires are reviewed and commented by 3 lactation consultants and 2 midwives and revised accordingly.
Change of breastfeeding self-efficacy (mothers' confidence in their abilities to breastfeed their babies) by the Chinese Hong Kong version of Breastfeeding Self-Efficacy Scale-Short Form (BSES-SF) from baseline to 6 months after delivery | At baseline, 2 months (immediately post-intervention) and 6 months postpartum
  BSES-SF is a 14-item scale with 5-point Likert scale. Total score ranged from 14 to 70 and higher score indicates higher breastfeeding self-efficacy. and the results will be presented as BSES-SF mean scores which are measured by Breastfeeding Self-Efficacy Scale-Short Form (BSES-SF) (Dennis, 2003)

SECONDARY OUTCOMES:
Partial breastfeeding rate (number of infants who have been fed with breastmilk together with formula milk or other food/ liquids) by self-developed postnatal questionnaires | At 2 months and 6 months postpartum
  The self-developed postnatal questionnaires are reviewed and commented by 3 lactation consultants and 2 midwives and revised accordingly.
Breastfeeding initiation rate (number of mothers initiate breastfeeding within 1st hour of delivery) by self-developed postnatal questionnaire | At 2 months postpartum
  The self-developed postnatal questionnaire are reviewed and commented by 3 lactation consultants and 2 midwives and revised accordingly.
Exclusive breastfeeding duration (total length of time on exclusive breastfeeding) by self-developed postnatal questionnaires | At 2 months and 6 months postpartum
  The self-developed postnatal questionnaire are reviewed and commented by 3 lactation consultants and 2 midwives and revised accordingly.
Maternal postnatal depression score by the Chinese version of Edinburgh Postnatal Depression Scale (EPDS) | At 2 months and 6 months postpartum
  Maternal postnatal depression is one kind of mood disorder, which commonly occurs after the birth of a baby.
  In EPDS, there are 10 questions with a total score of 0 to 30. Risk of postnatal depression was defined as EPDS score ≥10, and higher score indicates higher risk of a women suffering from postnatal depression.
Infant's morbidity (total number of infants getting sick and the types of infectious diseases that requires medical checkup) by self-developed postnatal questionnaires | At 2 months and 6 months postpartum
  The medical diseases to be estimated for these morbidities are limited to infectious diseases including respiratory, ear and gastrointestinal infection.
  The self-developed postnatal questionnaire are reviewed and commented by 3 lactation consultants and 2 midwives and revised accordingly.

CONTACTS AND LOCATIONS:
Locations (1):
- Natural Parenting Network, Hong Kong, Hong Kong

REFERENCES:
- [Derived] Wong MS, Chien WT. Effects of an Online Theory-Based Educational Programme for Primiparous Women on Improving Breastfeeding-Related Outcomes: A Randomised Controlled Trial. Scand J Caring Sci. 2025 Mar;39(1):e13320. doi: 10.1111/scs.13320. PMID 39865520
- [Derived] Wong MS, Chien WT. A Pilot Randomized Controlled Trial of an Online Educational Program for Primiparous Women to Improve Breastfeeding. J Hum Lact. 2023 Feb;39(1):107-118. doi: 10.1177/08903344221125129. Epub 2022 Oct 3. PMID 36189735